CLINICAL TRIAL: NCT02329158
Title: Clinical Impact of Disinvestment in Hydroxyl-ethyl Starches (HES) for Patients Undergoing Cardiac Surgery
Brief Title: Disinvestment in Hydroxyl-ethyl Starches (HES) for Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 105755
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Cardiac Surgical Procedures
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm: Exposed: Hydroxyethyl starch: Cardiac surgical patients exposed to 6% hydroxyethyl starch (130/0.4).
  Interventions: Drug: 6% hydroxyethyl starch
- Arm: Unexposed: Hydroxyethyl starch: Cardiac surgical patients not exposed to 6% hydroxyethyl starch (130/0.4).

INTERVENTIONS:
Drug: 6% hydroxyethyl starch
  Other Names: Voluven (Fresenius Kabi)
  Groups: Arm: Exposed: Hydroxyethyl starch

SUMMARY:
The purpose of this study is to determine whether disinvestment in hydroxyl-ethyl starches (HES) for patients undergoing cardiac surgery was safe and effective.

DETAILED DESCRIPTION:
Fluid replacement therapy is administered to patients requiring volume resuscitation following significant blood loss, or for maintenance fluid requirements. Severe blood loss can lead to anemia, reduced oxygen carrying capacity, and organ failure. Options for fluid replacement include red blood cell transfusion, colloids such as hydroxyethyl starches (HES), albumin, and gelatin as well as crystalloids such as normal saline and Ringer's lactate. Until recently, use of HES at the London hospitals and other major health sciences centers was concentrated in cardiac surgery patients and non-critically ill perioperative patients. In April 2013, the London Health Sciences Centre (LHSC) opted to discontinue the use of HES altogether, based on evidence suggesting that HES may be harmful compared to alternative fluid therapies.

The decision to disinvest in HES became effective on April 2, 2013. The hospitals no longer purchased HES, and clinicians used alternative fluids for volume resuscitation. Alternatives available at the hospitals included Ringer's lactate, normal saline, and albumin. All HES product was removed from patient care areas.

The investigators will perform a before/after analysis of the impact of HES disinvestment using a retrospective observational cohort study design, employing data obtained from administrative and clinical databases. Exposure to HES before disinvestment will be assumed to be 100% of cardiac surgical patients, and, after a washout period surrounding the time of disinvestment, exposure to HES will be assumed to be 0% after disinvestment.

The study population will be defined retrospectively in terms of the intervention received and the time period of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The London Health Sciences Centre disinvested in hydroxyethyl starches on April 2, 2013. The study population will include individuals undergoing cardiac surgery and discharged from hospital in one of two eras:

  * Era 1 (365 days prior to disinvestment in HES): the time period between April 1, 2012 and March 31, 2013, or
  * Era 2 (365 days following disinvestment in HES): the time period between June 1, 2013 and May 31, 2014 (NB: after a 2-month washout period to ensure all HES supplies had been exhausted).
* Specifically, the study population will be comprised of patients who underwent the following cardiac surgical procedures:

  * Coronary artery bypass graft only
  * Coronary artery bypass graft with aortic valve replacement
  * Coronary artery bypass graft with aortic valve repair
  * Coronary artery bypass graft with mitral valve replacement
  * Coronary artery bypass graft with mitral valve repair
  * Coronary artery bypass graft with a valve surgical procedure (replacement and/or repair) involving up two valves

Exclusion Criteria:

* Individuals undergoing heart transplants, aortic dissections, and other cardiac procedures not listed in the inclusion criteria above will be excluded.
* Individuals with any portion of the acute length of stay spanning the washout period (April 1, 2013 to May 31, 2013) will be excluded. Specifically, the following patients will be excluded:

  * Patients admitted prior to April 1, 2013 that remained in hospital on April 1, 2013.
  * Patients admitted during the washout period (April 1, 2013 to May 31, 2013) that remained in hospital on May 31, 2013.
  * Patients admitted and discharged during the washout period.
* We will exclude subsequent cardiac surgical procedures for individuals meeting the inclusion criteria more than once during the study timeframe (i.e. each patient's data will only be used once).
* Individuals enrolled in the randomized controlled clinical trial entitled, "VolulyteTM in Cardiac Surgery" (ClinicalTrials.gov Identifier: NCT01553617) will be excluded from the cohort. The purpose of this study was to assess the efficacy and safety of 6 % Hydroxyethyl Starch 130/0.4 in an Isotonic Electrolyte Solution (VolulyteTM) compared to 5% Human Serum Albumin as volume replacement therapy in elective open-heart surgery in adult patients on cardiopulmonary bypass. Individuals enrolled in the trial were randomized to priming of the cardiopulmonary bypass machine and volume therapy as necessary with either Volulyte or Human Serum Albumin. The study began in October 2012 and was completed in January 2014, with a total enrolment of 133 patients. The approximate number enrolled at LHSC was 30. Because the study period overlaps with that of the pre- and post- disinvestment eras, individuals enrolled in this study will be excluded from the retrospective cohort.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The proposed study population includes adult patients (age >/= 18) who underwent coronary artery bypass surgery (CABG) with or without valve surgery at the London Health Sciences Centre.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Length of Stay | Following cardiac surgery (on average approximately 10 days)
  Acute hospital length of stay (in days) following cardiac surgery

SECONDARY OUTCOMES:
Rates of transfusion | During or after cardiac surgery, prior to hospital discharge (on average approximately 10 days)
  The proportion receiving a transfusion of red blood cells or other products.
Rates of transfusion | During or after cardiac surgery, prior to hospital discharge (on average approximately 10 days)
  The number of units of red blood cells or other products transfused.
Kidney Injury | During or after cardiac surgery, prior to hospital discharge (on average approximately 10 days)
  The proportion experiencing kidney injury as measured by serum creatinine levels.
Renal Replacement Therapy | During or after cardiac surgery, prior to hospital discharge (on average approximately 10 days)
  The proportion receiving renal replacement therapy.
Cost of care | During the acute phase of the hospital stay (on average approximately 10 days)
  The total cost of the acute phase of hospitalization based on hospital case cost data.
In-hospital mortality | Death during the hospital stay (on average approximately 10 days)
  The proportion dying during the hospital stay.

REFERENCES:
- [Derived] Hong M, Jones PM, Martin J, Kiaii B, Arellano R, Cheng D, John-Baptiste AA. Clinical impact of disinvestment in hydroxyethyl starch for patients undergoing coronary artery bypass surgery: a retrospective observational study. Can J Anaesth. 2019 Jan;66(1):25-35. doi: 10.1007/s12630-018-1245-5. Epub 2018 Nov 8. PMID 30411246